CLINICAL TRIAL: NCT04103541
Title: Epigenetic Impact of a Psychotherapeutic Program in Adolescents With Severe Adverse Experiences
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2019-0189; Psychology, (Other: UW, Madison)
Record Dates: First submitted 2019-09-23; First posted 2019-09-25 (Actual); Last update posted 2019-09-26 (Actual); Status verified 2019-09

CONDITIONS: Children Exposed to Adverse Experiences

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- IP-Colombia (Experimental)
  Interventions: Behavioral: IP-Colombia
- Waitlist control (No Intervention)

INTERVENTIONS:
Behavioral: IP-Colombia — The IP-Colombia program is a multi-component intervention carried out in the context of therapeutic camp, based on EDMR therapies and mindfulness-based interventions. Alongside the interventions, activities are done to facilitate healthy lifestyles, empathy, [and] the recognition and expression of emotions through exercise, art workshops, musical creation, dance and theater.
  Arms: IP-Colombia

SUMMARY:
In this project, the investigator proposes to examine the influence of a psychotherapeutic program, designed for adolescents with a history of early adverse environmental and psychosocial experiences, on gene expression in order to find ways to reverse critical molecular mechanisms that associate extreme childhood stress with the development of a series of health problems, with important repercussions at both the individual and social levels.

DETAILED DESCRIPTION:
The investigator proposes a randomized controlled clinical trial to be attended by adolescents who are in the process of re-establishing their rights with the Colombian Family Welfare Institute. The study team will compare the genome methylation states of saliva samples from a group of 21 adolescents (children, ages 13 to 16), [both] before and after an 8-day residential intervention (IP-Colombia psychotherapeutic program). A randomized control group (waitlist) (n=21) will be included, from which baseline samples and samples after 8 days in their usual living conditions will be collected. For randomization, the evaluation of exposure to stress during childhood will be measured by using a questionnaire on adverse experiences.

The IP-Colombia program is a multi-component intervention carried out in the context of therapeutic camp, based on Eye Movement Desensitization and Reprocessing (EMDR) therapies and mindfulness-based interventions. Alongside the interventions, activities are done to facilitate healthy lifestyles, empathy, [and] the recognition and expression of emotions through exercise, art workshops, musical creation, dance and theater. Previous studies carried out by the Colombia Innocence in Danger Foundation have shown the significant effects of the IP-Colombia protocol in the treatment of children with post-traumatic stress disorder associated with severe interpersonal violence. The Colombia Innocence in Danger Foundation team, which has 10 years of experience with this intervention that has benefited around 380 boys, girls, and teenagers, will be responsible for this intervention.

The molecular analysis will be coordinated by Dr. Perla Kaliman, a collaborating researcher at the Center for Healthy Minds at the University of Wisconsin-Madison, directed by Dr. Richard Davidson. Dr. Kaliman, in collaboration with Dr. Davidson, has conducted the first studies showing the epigenetic effects of stress-reduction interventions. The DNA processing and methylome analysis will be carried out at the University of Wisconsin-Madison, in Dr. Reid Alisch's laboratory [by] a team recognized worldwide for its experience in the epigenetics of adverse experiences in young people.

The saliva samples will be collected in duplicate, using Oragene kits for DNA methylation analysis (DNA Genotek, Canada). The samples will be sent immediately after collection at room temperature to the Center for Healthy Minds (Madison, Wisconsin).

The DNA will be extracted using the Qiagen kit for human saliva samples, following the manufacturer's protocol. The genomic DNA samples will be analyzed in a 1% agarose gel, to verify that the DNA is of high molecular weight, and they will be quantified using Qubit (Qiagen, USA). DNA methylation levels will be determined using the HumanMethylation450 (Illumina) and the beta values will be obtained using the R min package. Methylation data that correspond to the methylation in a Single nucleotide polymorphism (SNP) will be eliminated from the analysis if they contain a SNP within the probe, if they are known to cross-react, or if a sample has a detection P-value > 0.01.

ELIGIBILITY:
Inclusion Criteria:

* Adolescents in the process of reestablishing their rights with the Colombian Family Welfare Institute.

Exclusion Criteria:

-

Ages: 13 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 44 (Actual)
Dates: Start 2019-06-01 (Actual); Primary Completion 2019-07-01 (Actual); Study Completion 2019-07-01 (Actual)

PRIMARY OUTCOMES:
Change in the level of DNA methylation following IEP-Colombia psychotheraupeutic program | Baseline and after day 8
  Saliva sample from children who were exposed to adverse experience during their childhood, will be examined for DNA methylation levels at roughly half a million sites. This will occur both before and after attending the Individualized Education Program(IEP)-Colombia psychotherapeutic program. Epigenetic modifications, such as DNA methylation, are mechanisms for regulating gene expression that are strongly influenced by environment, experiences, and lifestyle.

SECONDARY OUTCOMES:
Change in Short PTSD Rating Interview (SPRINT) score following IEP-Colombia psychotheraupeutic program | Baseline and after day 8
  SPRINT is an eight-item self-report measure that assesses the core symptoms of PTSD (intrusion, avoidance, numbing, arousal), somatic malaise, stress vulnerability, and role and social functional impairment. The SPRINT does not map onto any specific version of Diagnostic and Statistical Manual of Mental Disorders (DSM) but rather is intended to capture the common symptoms that tend to be reported by people with PTSD when first seeking care. SPRINT is responsive to symptom change over time and can serve as a measure of PTSD illness severity and of global improvement. Symptoms are rated on five-point scales from 0 (not at all) to 4 (very much) and the authors suggest a cutoff score of 14 for this screen. Those receiving positive scores should be further assessed.
Change in Mindful Attention and Awareness Scale for Adolescents (MAAS-A) score following IEP-Colombia psychotheraupeutic program | Baseline and after day 8
  The MAAS is a 15-item scale designed to assess a core characteristic of dispositional mindfulness, namely, open or receptive awareness of and attention to what is taking place in the present. The items are answered on a six-point scale (1=Almost always; 6=Almost never) on which higher scores are an indication of higher trait mindfulness.
  The scale shows strong psychometric properties and has been validated with college, community, and cancer patient samples. Correlational, quasi-experimental, and laboratory studies have shown that the MAAS taps a unique quality of consciousness that is related to, and predictive of, a variety of self-regulation and well-being constructs. The measure takes 10 minutes or less to complete.

OTHER OUTCOMES:
Assessment of Childhood Adverse Experiences (ACEs). | At Baseline
  The Adverse Childhood Experience (ACE) Questionnaire is a 10-item self-report measure developed for the ACE study to identify childhood experiences of abuse and neglect. The survey consists of ten questions. Each affirmative answer is assigned one point. At the end of the questionnaire, the points are totaled for a score out of ten, which is known as the ACE score.
  ACEs at baseline may be used as co-variate measure.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Wisconsin Madison, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No
All data received by the Center for Healthy Minds will be coded. These data will be stored on dedicated servers, housed in a data center with access limited to authorized personnel. "Although not fully described in this application, any future research using this study data will remain in line with the original study's objectives and themes." "Specimens will not be returned to the lead site. They will be destroyed after analysis."
  Hard copies of study materials, such as consent forms and screening logs, will remain at Universidad de Santander, as will the key that links identifiable information to coded data.
  Access to study data is restricted to lab computers by the use of a network firewall, and further restricted only to users specifically authorized for each study. Access to data is disabled when a user leaves the lab. Periodic audits verify system integrity and security, and account activity.